CLINICAL TRIAL: NCT01473719
Title: Reducing STIs in Emerging Adults Who Use Alcohol and Marijuana
Brief Title: Emerging Adults Who Use Alcohol and Marijuana
Acronym: HEAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Principal Investigator, Michael Stein, MD, Principal Investigator, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AA020509 (NIH)
Record Dates: First submitted 2011-11-15; First posted 2011-11-17 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Alcohol Use; Marijuana Use; Sexually Transmitted Infections
Keywords: alcohol use; marijuana use; STI
MeSH Terms: conditions — Alcohol Drinking; Marijuana Use; Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- motivational intervention (Active Comparator): 7-session individual motivationally-based intervention
  Interventions: Behavioral: motivational intervention
- health education (Placebo Comparator): 7-session individual session focusing on health education
  Interventions: Behavioral: health education

INTERVENTIONS:
Behavioral: motivational intervention — 7-session individual motivationally-based intervention
  Arms: motivational intervention
Behavioral: health education — 7 individual sessions focusing on health education
  Arms: health education

SUMMARY:
The purpose of this study is to if a brief motivational intervention, compared to health education sessions, reduces alcohol and marijuana use and is related to fewer sexually transmitted infections (STI)in emerging adults who are engaging in alcohol and marijuana use.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 25
* Binge drink (5 or more drinks in a 2-hour period for men, 4 or more for women) at least monthly
* Use marijuana at least weekly
* Have been heterosexually active in the past six months
* Are not married
* Have not been living with a sexual or romantic partner for more than 6 months
* Be English speaking
* Reside within 20 miles of Providence, RI and plans to stay in the geographic area for the next 15 months
* Provide contact information for at least two verifiable locator persons

Exclusion Criteria:

* Have DSM-IV diagnosis of drug abuse or dependence (other than nicotine, marijuana)
* Have DSM-IV diagnosis of alcohol dependence

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 566 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
alcohol use | 15 months
marijuana use | 15 months
sexually transmitted infection | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Stein, MD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Caviness CM, Anderson BJ, Stein MD. Impact of Nicotine and Other Stimulants on Sleep in Young Adults. J Addict Med. 2019 May/Jun;13(3):209-214. doi: 10.1097/ADM.0000000000000481. PMID 30461442
- [Derived] Caviness CM, Anderson BJ, Stein MD. Energy drinks and alcohol-related risk among young adults. Subst Abus. 2017 Oct-Dec;38(4):376-381. doi: 10.1080/08897077.2017.1343217. Epub 2017 Jun 16. PMID 28622099
- [Derived] Moitra E, Christopher PP, Anderson BJ, Stein MD. Coping-motivated marijuana use correlates with DSM-5 cannabis use disorder and psychological distress among emerging adults. Psychol Addict Behav. 2015 Sep;29(3):627-32. doi: 10.1037/adb0000083. Epub 2015 Apr 27. PMID 25915689
- [Derived] Caviness CM, Tzilos G, Anderson BJ, Stein MD. Synthetic Cannabinoids: Use and Predictors in a Community Sample of Young Adults. Subst Abus. 2015;36(3):368-73. doi: 10.1080/08897077.2014.959151. Epub 2014 Sep 15. PMID 25222129